CLINICAL TRIAL: NCT00638053
Title: Head Trauma With Traumatic Brain Injury (TBI): A Multicenter, Phase IV Study to Evaluate the Effects of Genotropin in Adult Patients With Growth Hormone Deficiency (GHD) Caused by Trauma and/or Head Injury
Brief Title: A Study to Evaluate the Efficacy of Somatropin in Adults With Growth Hormone Deficiency Caused by Trauma and/or Head Injury
Acronym: GHD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See reason for termination in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GENGHD-0018-078
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Brain Injuries; Growth Hormone Deficiency Dwarfism
MeSH Terms: conditions — Brain Injuries; Dwarfism, Pituitary | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Genetic: somatropin

INTERVENTIONS:
Genetic: somatropin — Somatropin will be administered as a daily subcutaneous injection; Fixed doses starting with 0.1 mg/day in patients older than 55 years or patients weighing less than 50 kg; all other patients: 0.1 mg/day or 0.2 mg/day (these doses should all be lower than 0.04 mg/kg/week); all patients starting at 0.1 mg/day will have their dose progressively increased in 0.1 mg/day increments to a maximum clinically- and pharmacologically- tolerated plateau dose; all patients starting at 0.2 mg/day will increase in 0.2 mg/day increments; all incremented dose changes will occur at monthly intervals based on IGF-I levels; treatment will continue for 12 months

SUMMARY:
The purpose of this study is to assess the prevalence of GHD in patients who sustain a head injury or suffer a major traumatic event and to evaluate the efficacy of growth hormone (GH) therapy in the treatment of GHD caused by trauma or head injury

DETAILED DESCRIPTION:
The study was terminated on October 9, 2003. The reason cited for the termination was due to poor patient recruitment and therefore not enough data could be collected to provide comprehensive analysis for reporting of results. No safety or efficacy issues were reported to cause the termination of the study.

ELIGIBILITY:
Inclusion Criteria:

* Documented GHD
* Documented mild, moderate, and severe head injury (e.g.,Glasgow COMA Scale score less than or equal to 15 or equivalent measure)

Exclusion Criteria:

* Active systemic malignancy or active intracranial tumor
* Growth hormone replacement therapy in the last 12 months
* History of dementia unrelated to traumatic brain injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2002-11; Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Change in the serum Insulin-like growth factor-I (IGF-I)concentration from baseline | Months 1 thru 11
Number of patients with abnormal GH stimulation tests | Baseline

SECONDARY OUTCOMES:
Change from baseline in waist circumference | Month 12
Age and gender specific optimal doses of GH replacement | Months 1 thru 11
Change in Quality of Life-Adult Growth Hormone Deficiency Assessment | Months 1 thru 12
Assessment of adverse events | Months 1 thru 12
Serum prolactin, thyroid stimulating hormone, free thyroxine serum, cortisol, adrenocorticotropic hormone, luteinizing hormone, follicle stimulating hormone, estradiol, and testosterone to assess degree of other anterior pituitary hormone deficiencies | Baseline
Change from baseline in Glasgow Outcome Score | Month 12
Change in Quality of Life-Mini-Mental scores | Months 1 thru 12

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Federal Way, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=GENGHD-0018-078&StudyName=A%20Study%20to%20Evaluate%20the%20Efficacy%20of%20Somatropin%20in%20Adults%20with%20Growth%20Hormone%20Deficiency%20Caused%20by%20Trauma%20and/or%20Head%20Injury%20